CLINICAL TRIAL: NCT01285297
Title: A Prospective, Multicenter, Single Arm Study of Transmyocardial Revascularization (TMR) Plus Bone Marrow Aspirate Concentrated (BMAC) Using the Cardiogenesis PHOENIX Combination Handpiece Delivery System
Brief Title: Safety Study of Transmyocardial Revascularization (TMR) With Bone Marrow Aspirate (BMAC) for Angina Reduction
Acronym: PHOENIX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiogenesis Corporation, a wholly-owned subsidiary of CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX 09-003
Record Dates: First submitted 2010-12-14; First posted 2011-01-28 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Angina
Keywords: Transmyocardial revascularization (TMR); Bone marrow aspirate concentrate (BMAC); Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMR plus BMAC injection (Experimental): Injection of bone marrow aspirate concentrate into reversibly ischemic myocardium with transmyocardial revascularization during the same open procedure.
  Interventions: Biological: Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Biological: Bone Marrow Aspirate Concentrate — Injection of up to 18 mL BMAC

SUMMARY:
The purpose of this study is to determine the safety of injecting autologous bone marrow concentrate with laser transmyocardial revascularization (TMR) for treatment of angina which cannot be treated by direct coronary intervention.

DETAILED DESCRIPTION:
Recently published information suggests the delivery of concentrated autologous bone marrow, in combination with transmyocardial revascularization (TMR) may provide synergistic effects for the reduction of angina in patients who are not treatable with conventional coronary artery bypass or percutaneous coronary intervention. This safety and feasibility study is intended to confirm the work previously done at one hospital in a larger, multicenter setting. Patients who are candidates for TMR will be asked to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, 18 years of age or older, male or female.
* Left ventricular ejection fraction greater than or equal to 40% (documented within 6 months of the TMR procedure.
* Patient with medically refractory, stable, Class IV angina according to the Canadian Cardiovascular Society angina scale. Optimal medical therapy is defined as maximum tolerable and stable doses of beta-blockers, statins, anti-platelets and long acting nitrates without control of symptoms for at least 30 days.
* Patient with at least a 15 cm² (or 15% of the surface area in the distal 2/3 of the left ventricle free wall to allow for a minimum of 15 TMR channels) documented region of the myocardium in the distal two-thirds of the left ventricle with reversible ischemia. Patients will be enrolled based on images used to determine eligibility for TMR within the previous 6 months. However, all patients will have baseline and follow-up MRIs taken per a standardized protocol and adjudicated by a core lab.
* Has a documented left ventricular wall thickness of ≥8 mm.
* Patient is not a candidate for treatment by direct coronary revascularization methods (i.e., CABG or PCI) as documented by an independent interventional cardiologist and an independent cardiothoracic surgeon on the Angiographic Screening Form.
* Patient is able to perform the baseline exercise tolerance test (ETT).
* Patient, if female, has no childbearing potential or has had a negative urine or serum pregnancy test within 7 days of the procedure.
* Patient has a bone marrow aspirate total nucleated count of at least 15 x 106/mL at the time of harvest.
* Patient has provided informed consent.

Exclusion Criteria:

* Cannot undergo a surgical procedure, thoracotomy or general anesthesia.
* Has any mechanical or prosthetic heart valve.
* Has a history of bone marrow disease (especially Non-Hodgkin's Lymphoma and Myelodysplastic Syndrome) that prohibits autologous bone marrow derived cell transplantation.
* Has severe, new onset or increasing angina. In addition, patients who cannot be weaned from intravenous anti-anginal medications for at least 48 hours preoperatively are to be excluded. Severe, new onset and increasing angina is defined as: Severe angina - angina occurring at rest and usually prolonged >20 minutes occurring within a week of presentation; new onset angina - angina of at least Canadian Cardiovascular Society Classification (CCSC) III severity with onset within 2 months of initial presentation; and increasing angina - previously diagnosed angina that is distinctly more frequent, longer in duration, or lower in threshold, (i.e., increased by at least one CCSC class within 2 months of initial presentation to at least CCSC III severity.
* Has had a STEMI (ST Elevation Myocardial Infarction) or NSTEMI (Non-STEMI) within 4 weeks of the TMR procedure.
* Has decompensated heart failure, or a diagnosis of NYHA Functional Class III/IV heart failure.
* Has a hemorrhagic propensity that cannot be addressed with drug management.
* Has severe or life-threatening arrhythmia (e.g., ventricular tachycardia or fibrillation) within one week prior to the TMR procedure.
* Is unable to undergo a cardiac MRI procedure.
* Has uncontrolled diabetes with HbA1C > 10%.
* Has anemia defined as hematocrit < 33% in women and <39% in men.
* Has moderate to severe renal dysfunction defined as serum creatinine >1.8 mg/dL.
* Has moderate to severe liver dysfunction defined as> ALT/AST >5X the upper limit of normal.
* Is unable or unwilling to return for follow-up.
* Is participating in another clinical investigation within the prior 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events (MACCE) | One Year
  MACCE is defined as cardiac death, cerebrovascular accidents, myocardial infarction, serious arrhythmia and congestive heart failure
Mortality | One Year
  All cause mortality

SECONDARY OUTCOMES:
Exercise Tolerance Test | 3, 6 and 12 months
  Exercise tolerance to onset of moderately severe angina
Ejection Fraction | 6 and 12 months
  Ejection fraction and areas of myocardial ischemia by cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Keith B Allen, MD, Study Director — Clinical Advisor
Locations (2):
- Bakoulev Scientific Center for Cardio-vascular Surgery, Moscow, Russia
- Hospital Universitario de La Princesa, Madrid, Spain

REFERENCES:
- [Background] Reyes G, Allen KB, Aguado B, Duarte J. Bone marrow laser revascularisation for treating refractory angina due to diffuse coronary heart disease. Eur J Cardiothorac Surg. 2009 Jul;36(1):192-4. doi: 10.1016/j.ejcts.2009.03.022. Epub 2009 Apr 25. PMID 19394846